CLINICAL TRIAL: NCT07093190
Title: Effect of Rg1 Supplementation on Stem Cells in Exercised Skeletal Muscles of Women > 60 y
Brief Title: Stem Cell Recruitment in Exercised Skeletal Muscles of Older Women by Phytosteroid Rg1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Taipei (Other)
Responsible Party: Principal Investigator, Chia-Hua Kuo, Professor, University of Taipei
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB-2021-045; NSTC 110-2622-H-845-004 (Other Grant/Funding Number: National Science Technology Council Taiwan-Nuliv Science USA); 13A1-CG-CO-05-2426-3 (Other Grant/Funding Number: National Health Research Institutes (Taiwan))
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Exercise Training; Post-menopausal Women; Bone Marrow Stem Cells; Skeletal Muscle Recovery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise following Rg1 consumption (Experimental): 1 hour following the consumption of the Rg1 supplement, participants performed exercise intervention before muscle biopsies were taken.
  Interventions: Dietary Supplement: exercise following Rg1 consumption
- exercise only following placebo consumption (Placebo Comparator): Crossover trial with placebo supplementation consumed before exercise
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: exercise following Rg1 consumption — The effect of Rg1 on exercised skeletal muscle in older women
  Arms: exercise following Rg1 consumption
Dietary Supplement: Placebo — Resistance exercise performed 1 hour following placebo consumption
  Arms: exercise only following placebo consumption

SUMMARY:
The goal of this interventional study is to observe the effects of bone marrow stem cell behavior in skeletal muscle of women between 60 to 75 years old after a single moderate resistance exercise session. Plant sterol Rg1, a compound known to enhance stem cell infiltration following exercise in young men will be tested against a placebo in a double blinded crossover design.

The main questions to be answered are:

* Does Rg1 supplementation alter serum sex hormone levels in recovery from exercise?
* Does Rg1 supplementation influence bone marrow stem cell differentiation in skeletal muscles of older women?

Participants will:

* Pre-test body composition, maximal leg strength, blood and muscle tissue.
* One hour after taking the supplement, participants will perform 4 sets of 10 repetitions of 70% of maximal strength (1RM) leg press and have two thigh muscle biopsies (0 and 24 h after exercise).
* Repeat the protocol one month later on the alternative supplement. Researchers will understand whether Rg1 improves recovery response to resistance exercise in post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* sedentary, able to cease medications and supplements for 48 h before and 24 h after exercise session, medically sound for lower body moderate resistance exercise

Exclusion Criteria:

* use of insulin, sex hormone and immune-modulating medications, smoking and regular alcohol consumption

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Stro-1+ bone marrow stem cell area in skeletal muscle biopsies | from enrolment to the end of study at 8 weeks
  Immunofluorescence staining will be used to semi-quantitatively analyze Stro-1+ BMSC presence in skeletal muscle of older women before, 0h and 24h after a moderate resistance exercise session.
Nestin+ neural stem cell area in skeletal muscle biopsies | from enrolment to the end of study at 8 weeks
  Immunofluorescence staining will be used to semi-quantitatively analyze Nestin+ neural stem cell presence in skeletal muscle of older women before, 0h and 24h after a moderate resistance exercise session.
CD34+/CD31+ vascular stem cell area in skeletal muscle biopsies | from enrolment to the end of study at 8 weeks
  Immunofluorescence staining will be used to semi-quantitatively analyzeCD34+/CD31+ vascular stem cell presence in skeletal muscle of older women before, 0h and 24h after a moderate resistance exercise session.
Serum sex hormone levels 24 h following resistance exercise | from enrolment to the end of study at 8 weeks
  Forearm blood draw and Elisa analysis of serum for estradiol, progesterone, and testosterone of older women before and 24h after a moderate resistance exercise session.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-hua Kuo, PhD, Principal Investigator — University of Taipei
Locations (1):
- University of Taipei, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The National Research Institutes of Health (Taiwan) will conduct gene analysis on remaining muscle samples for aiding understanding of sarcopenia

REFERENCES:
- [Background] Glaziou P, Martin PM. Study of factors that influence the clinical response to ciguatera fish poisoning. Toxicon. 1993 Sep;31(9):1151-4. doi: 10.1016/0041-0101(93)90130-b. PMID 8266347